CLINICAL TRIAL: NCT06084312
Title: Contact Registry for Clinical Trials At the University of Central Florida College of Medicine
Brief Title: Contact Registry for Clinical Trials
Status: Recruiting | Type: Observational
Sponsor: University of Central Florida (Other)
Responsible Party: Sponsor
Other Study IDs: STUDY00004132
Record Dates: First submitted 2023-10-03; First posted 2023-10-16 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: This is the Contact Registry
Keywords: Healthy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 50 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- This registry will not target any specific populations

SUMMARY:
The purpose of the Contact Registry for Clinical Trials is to develop a database/listserv of persons interested in clinical trials occurring at the University of Central Florida College of Medicine.

Sign up for the UCF College of Medicine's Contact Registry for Clinical Trials to learn about clinical research and clinical trials in areas of interest to you!

https://ucf.qualtrics.com/jfe/form/SV_do4WGvKlz4f8Wwe

DETAILED DESCRIPTION:
The Contact Registry for Clinical Trials allow persons to sign up to learn more about clinical trials and clinical research around certain medical indications that will be occurring at the University of Central Florida College of Medicine. Persons are not asked to provide any personal health information. Persons are asked to provide identifying information needed to provide the requested information.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Persons who do not read English could register through the assistance of their friends or software for translation

Exclusion Criteria:

* Children may not register
* Persons who are unable to consent may not register

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This registry will not target any specific populations.
Sampling Method: Non-Probability Sample
Enrollment: 50000 (Estimated)
Dates: Start 2022-04-18 (Actual); Primary Completion 2030-01 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
To allow persons to sign up to learn more about clinical trials and clinical research around certain medical indications that will be occurring at the University of Central Florida College of Medicine | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- University of Central Florida, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No